CLINICAL TRIAL: NCT07403890
Title: Rewiring the Brain-Immune Axis for Chronic Pain Using Transcranial Magnetic Stimulation in Psoriatic Arthritis
Acronym: REACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GN25RH492
Record Dates: First submitted 2026-01-16; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: Participants are randomised 1:1 to receive either active rTMS to the left inferior parietal lobule or control rTMS to the vertex for 12 sessions over 4 weeks.
Who Masked: Participant
Masking Description: Participants are masked to group allocation. The rTMS operator is not masked due to the need to position the coil at different stimulation sites.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (Left Inferior Parietal Lobule) (Experimental): Participants receive active repetitive transcranial magnetic stimulation (rTMS) targeted to the left inferior parietal lobule (L-IPL). Stimulation is delivered at 10 Hz, 90% resting motor threshold, 1200 pulses per session, across 12 sessions over 4 weeks. This arm is designed to evaluate whether neuromodulation of the L-IPL alters immune signalling and reduces persistent pain in psoriatic arthritis.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS)
- rTMS (Vertex Stimulation) (Sham Comparator): Participants receive control rTMS delivered to the cranial vertex, a site not expected to modulate neuroimmune pathways relevant to pain. Stimulation parameters match the active arm (10 Hz, 90% resting motor threshold, 1200 pulses per session, 12 sessions over 4 weeks). This arm controls for nonspecific effects of rTMS, including sensory experience and participant expectations.
  Interventions: Device: Control Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS delivered to the left inferior parietal lobule at 10 Hz, 90% resting motor threshold, 1200 pulses per session, for 12 sessions over 4 weeks.
  Arms: rTMS (Left Inferior Parietal Lobule)
Device: Control Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS delivered to the cranial vertex using identical stimulation parameters to the active arm, serving as a control condition.
  Arms: rTMS (Vertex Stimulation)

SUMMARY:
Despite advances in immunomodulatory therapies, many Psoriatic arthritis (PsA) patients experience persistent pain unrelated to clinical active joint inflammation. Recent evidence suggests the Inferior Parietal Lobule (IPL) serves as a neuroimmune hub linking central neural activity with peripheral immune dysregulation. In a prior feasibility study, a single L-IPL-targeted TMS session reduced pain and altered immune signalling in inflammatory arthritis by reducing STAT3 phosphorylation in circulating monocytes. This study builds on those findings by evaluating whether rTMS over 4 weeks can induce sustained immune reprogramming while providing meaningful pain relief.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic immune-mediated inflammatory disease (IMID) characterised by musculoskeletal pain, enthesitis, and synovitis. While advances in immunomodulatory therapies have improved control of inflammation, approximately one-third of people with PsA continue to report persistent pain despite achieving low disease activity by clinical criteria. This dissociation between detectable inflammation and ongoing pain suggests a role for central nervous system (CNS) mechanisms in the persistence of symptoms. Emerging evidence from neuroimaging studies has highlighted the inferior parietal lobule (IPL) as a brain region implicated in both pain perception and immune signalling. Prior work in inflammatory arthritis shows that IPL grey-matter volume and functional connectivity correlate with peripheral inflammation and pain.

These findings suggest that the IPL may act as a neuroimmune hub, integrating nociceptive input and modulating pain perception and immune function via top-down signalling pathways. Recent translational research across cancer, cardiovascular, and IMIDs has established that brain activity can shape peripheral immune responses, and thereby influence disease progression.

In PsA, chronic pain may therefore reflect not only residual joint pathology but also maladaptive brain immune interactions that perpetuate inflammation and amplify pain processing. This under-explored pathophysiological loop constitutes a critical unmet therapeutic target in PsA and other IMIDs.

Psoriatic arthritis-related pain is only partially explained by joint specific inflammation. Despite excellent control of peripheral inflammation by contemporary immune modulatory regimes, as many as 30% of patients continue to report disabling levels of pain, thus comprising an urgent unmet clinical need.

Our group has been among the first to evidence a contributory role of the CNS as an explanation for this debilitating symptom. Neuroimaging studies in inflammatory arthritis have highlighted the inferior parietal lobule (IPL) as a potential neuroimmune hub: altered IPL grey-matter volume and functional connectivity have been linked to both systemic inflammation and pain, suggesting this region may integrate nociceptive and immune signals. These findings are consistent with broader evidence implicating IPL hyperconnectivity in pro-nociceptive brain networks observed in chronic pain conditions such as fibromyalgia.

The investigators therefore propose that in PsA, the IPL acts as a key interface between the CNS and the immune system, contributing to persistent pain via maladaptive neuroimmune signalling. A recent feasibility study (Pro-BEPP) conducted by the investigative team provided preliminary support for this mechanism, demonstrating that a single session of L-IPL-targeted TMS reduced pain and modulated immune activity, specifically decreasing STAT3 phosphorylation in circulating monocytes. These findings support a novel model of top-down immune regulation, wherein modulation of brain activity reprograms systemic inflammatory responses.

Given the neuroplasticity of pain networks and the immunological relevance of monocytes and CD8⁺ T cells in PsA pathogenesis, the investigators hypothesise that rTMS targeting the L-IPL (an approach already approved in the NHS for treatment-resistant depression), can induce sustained immune adaptation and provide clinically meaningful pain relief. By combining neuromodulation with immune profiling, this study aims to generate mechanistic feasibility data to establish rTMS as a biologically grounded, non-pharmacological intervention for persistent pain in PsA.

The investigators hypothesise that the L-IPL functions as a neuroimmune interface in PsA, contributing to persistent pain via maladaptive signalling between the brain and the immune system. Specifically, the investigators propose that ongoing IPL hyperactivity and altered connectivity with pain-related networks contribute to heightened pain perception, even when peripheral inflammation appears well-controlled. This brain-immune dysregulation may further sustain or amplify systemic inflammation through top-down modulation of immune cells such as monocytes and CD8⁺ T cells, which are known to play key roles in PsA pathogenesis.

If this model is correct, then rTMS targeted to the left IPL will rebalance brain network activity and induce downstream changes in immune cell signalling, particularly reducing pro-inflammatory markers (e.g. STAT3 phosphorylation). The investigators expect this to translate into measurable improvements in pain and related symptoms, such as fatigue, representing a novel neuromodulatory approach for addressing persistent pain in PsA.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years ≤ 75 years
* Diagnosis of PsA according to CASPAR (Classification Criteria for Psoriatic Arthritis).
* Low disease activity (no more than one joint with clinically active swelling) or remission
* Chronic pain for at least 3 months and VAS (Visual Analogue Scale) pain ≥30 mm
* Stable treatment ≥3 months prior to entering the study
* Able and willing to maintain medication for the duration study
* Able to undergo MRI and TMS procedures

Exclusion Criteria:

* Inability to provide written informed consent.
* Severe physical impairment (e.g. blindness, deafness, paraplegia) Pregnant, planning pregnancy or breast feeding.
* Severe claustrophobia precluding MRI.
* Contraindications to MRI (e.g. metal implants/ pacemaker).
* Contraindications to TMS (e.g. history of seizures).
* Serious infection including sepsis, tuberculosis and opportunistic infections such as invasive fungal infections.
* Major confounding neurological disease including Multiple
* Sclerosis, Stroke, Traumatic Brain Injury, Parkinson's Disease, Alzheimer's Disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in STAT3 phosphorylation in circulating monocytes | Week 1 to Week 4
  Assessment of the effect of left-inferior parietal lobule (L-IPL) targeted repetitive transcranial magnetic stimulation (rTMS) on immune systems; specifically changes in circulating monocytes intracellular signalling, primarily STAT3 phosphorylation levels, assessed via flow cytometry, before and after rTMS targeting L-IPL compared with the control (vertex stimulation) condition.

SECONDARY OUTCOMES:
Changes in genetic expression of circulating immune cells, monocytes and CD8+ T-cells, using transcriptomic assays (RNA-seq). | Week 1 to Week 4
  Change in transcriptomic signatures of circulating monocytes and CD8⁺ T-cells, measured using RNA-sequencing to evaluate treatment-related alterations in immune cell gene expression.
Changes in trained immunity set-points in monocytes and CD8+ T-cells, by investigating their epigenetic profile changes using Cleavage Under Targets and Tagmentation (CUT&TAG assay). | Week 1 to Week 4
  Changes in trained immunity set-points within circulating monocytes and CD8+T-cells, investigated by epigenetic profiling using using Cleavage Under Targets and Tagmentation (CUT&Tag).
Changes in pain severity as measured by the Pain Number Rating Scale. | Week 1 to Week 4
  Change in pain severity assessed using the Numeric Rating Scale (0-10), where 0 indicates no pain and 10 indicates the worst pain imaginable.
Changes in pain severity as measured by Widespread Pain as part of the American College of Rheumatology Fibromyalgia scale. | Week 1 to Week 4
  Change in pain severity assessed using the Widespread Pain Index (0-19) from the American College of Rheumatology Fibromyalgia criteria, with higher scores indicating pain in a greater number of body regions.
Changes in putative pain confounders as measured by PROMIS-Fatigue. | Week 1 to Week 4
  Change in fatigue severity measured using the Patient-Reported Outcomes Measurement Information System - Fatigue (PROMIS-Fatigue) scale, reported as standardized T-scores (mean 50, SD 10), where higher scores indicate greater fatigue and lower scores reflect less fatigue
Changes in putative pain confounders as measured by PROMIS-Depression. | Week 1 to Week 4
  Change in depressive symptoms measured using the Patient-Reported Outcomes Measurement Information System - Depression (PROMIS-Depression) scale, reported as standardized T-scores (mean 50, SD 10), where higher scores indicate greater severity of depressive symptoms.
Changes in putative pain confounders as measured by PROMIS-Sleep Related Impairment. | Week 1 to Week 4
  Change in sleep-related impairment measured using the Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment (PROMIS- Sleep related impairment) scale, reported as standardized T-scores (mean 50, SD 10), with higher scores reflecting greater sleep disturbance and functional impairment due to poor sleep.
Changes in putative pain confounders as measured by PROMIS-Physical functioning short form. | Week 1 to Week 4
  Change in physical functioning measured using the Patient-Reported Outcomes Measurement Information System - Physical Functioning (PROMIS Physical Functioning) scale, reported as standardized T-scores (mean 50, SD 10). Higher scores indicate better physical functioning, while lower scores reflect greater functional limitation.
Changes in putative pain confounders as measured by PROMIS-Pain Interference. | Week 1 to Week 4
  Change in pain-related functional interference measured using the Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS Pain Interference) scale, reported as standardized T-scores (mean 50, SD 10), where higher scores indicate greater interference of pain with daily activities.
Changes in PsA disease activity as measured by Disease Activity in Psoriatic Arthritis (DAPSA). | Week 0 to Week 4
  Change in psoriatic arthritis disease activity measured using the Disease Activity in Psoriatic Arthritis (DAPSA) score, a composite index incorporating tender and swollen joint counts, patient pain, patient global assessment, and C-reactive protein. Higher scores indicate greater disease activity. Standard disease-activity categories are: remission (≤4), low (>4-14), moderate (>14-28), and high (>28).
Changes in PsA disease activity as measured by Minimal Disease Activity (MDA). | Week 0 to Week 4
  Change in psoriatic arthritis disease activity assessed using the Minimal Disease Activity (MDA) criteria, a composite measure based on seven domains (tender joint count, swollen joint count, patient pain, patient global assessment, skin involvement, enthesitis, and physical function). Participants are classified as achieving MDA when they meet at least five of the seven criteria.
Changes in PsA disease activity as measured by Body Surface Area (BSA). | Week 0 to Week 4
  Change in psoriatic disease activity assessed using Body Surface Area (BSA), which quantifies the percentage of skin affected by psoriasis, with higher values indicating greater disease involvement.
Changes in blood protein levels of inflammatory cytokines/chemokines. | Week 1 to Week 4
  Change in circulating protein levels of inflammatory cytokines and chemokines measured from blood samples collected at baseline and weekly throughout the intervention, to assess treatment-related alterations in systemic inflammatory signalling.

OTHER OUTCOMES:
Feasibility data on EQ-5D quality of life scores. | Week 1 and Week 4
  Feasibility of collecting EuroQol-5D-5L Questionnaire quality-of-life data assessed by the proportion of participants who complete the EQ-5D questionnaire at required study visits.
  The EQ-5D-5L includes five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels of severity, converted into a single index score ranging from below 0 to 1.0, where higher scores indicate better health-related quality of life.
Feasibility data on participant adherence. | Week 0 to Week 4
  Feasibility of participant adherence assessed by the proportion of scheduled rTMS visits attended across the 4-week intervention period, including adherence to interim assessments such as questionnaires and 7-day pain diaries.
Feasibility data on TMS tolerability. | Week 1 to Week 4
  Feasibility of TMS tolerability assessed by the frequency and severity of TMS-related adverse events recorded at each study visit across the 4-week intervention period.
Feasibility data on protocol completion rates. | Week 0 to Week 4
  Feasibility of protocol completion assessed by the proportion of participants who complete the 4-week intervention, defined as attending the required rTMS sessions (up to two allowable missed visits) and completing key study assessments (questionnaires, blood sampling, and MRI).
Neuroimaging biomarker: Left inferior parietal lobule to default mode network functional connectivity | Week 1 to Week 4
  Evaluation of how functional connectivity between the left inferior parietal lobule and the default mode network relates to treatment-associated changes in pain severity and immune markers, using resting-state functional magnetic resonance imaging to identify neuroimaging correlates of clinical and immunological improvement.
Neuroimaging biomarker: Left inferior parietal lobule to salience network functional connectivity | Week 1 to Week 4
  Evaluation of how functional connectivity between the left inferior parietal lobule and the salience network relates to treatment-associated changes in pain severity and immune markers, using resting-state functional magnetic resonance imaging to identify neuroimaging correlates of clinical and immunological improvement.
Neuroimaging biomarker: Left inferior parietal lobule to insula functional connectivity | Week 1 to Week 4
  Evaluation of how functional connectivity between the left inferior parietal lobule and the insula relates to treatment-associated changes in pain severity and immune markers, using resting-state functional magnetic resonance imaging to identify neuroimaging correlates of clinical and immunological improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Sunzini, MD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom